CLINICAL TRIAL: NCT00286416
Title: Double Blind Study to Determine Effect of Omalizumab Treatment in Patients With the Co-Morbid Conditions of Aspirin Exacerbated Respiratory Disease(AERD) and Allergic Asthma and Rhinitis.
Brief Title: Effect of Omalizumab (Xolair) in Treatment of Patients With AERD and Allergy Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scripps Clinic (Other)
Organization: Scripps Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Xolair AERD
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2006-01

CONDITIONS: Asthma; Allergic Rhinitis
Keywords: AERD; aspirin; allergy; omalizumab
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Hypersensitivity | interventions — Omalizumab

INTERVENTIONS:
Drug: omalizumab (Xolair)

SUMMARY:
Double blind protocol treatment of 2/3 of the patients with omalizumab and 1/3 placebo administer for 4 months. Patients selected for the study must have both aspirin exacerbated respiratory disease and allergic asthma and rhinitis. They must also have completed aspirin desensitization and be taking aspirin on a daily basis for the treatment of AERD.

DETAILED DESCRIPTION:
60 patients with Aspirin Exacerbated respiratory Disease will be screened to determine if they also have allergic respiratory tract disease as a co-morbid complication. This will involve history, allergy skin tests and a serum IgE level. They must also have been desensitized to aspirin and be taking aspirin 325 or 650 mg morning and night.

40/60 patients will receive omalizumab injections every month for the next 4 months and the other 20 patients, via a random program, will receive placebo injections.

Monthly visits with the nurse co-ordinator will involve the following assessments: daily symptom scores, daily use of medications (particularly prednisone and rescue albuterol inhalers), lung function tests, nasal breathing test, measurement of smell and quality of life scores pre and post study.

ELIGIBILITY:
Inclusion Criteria:

aspirin exacerbated respiratory disease and allergic asthma

Exclusion Criteria:

* pregnant females,starting immunotherapy in the past 3 months, prior treatment with Xolair, negative allergy skin tests,unable to participate in lung function tests, unable to complete data forms,low platelets, serum IGE greater than 700 iu,cancer,another uncontrolled medical condition, unacceptable concomitant medication, under the age of 18 years.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-01; Study Completion 2008-07

PRIMARY OUTCOMES:
Respiratory Index scores

SECONDARY OUTCOMES:
FEV1
Nasal Flow rates
Nasal smell scores
Quality of Life Scores for rhinitis and asthma

CONTACTS AND LOCATIONS:
Overall Officials: Gary Willaims, MD, PhD, Study Chair — Vice Chairman of Academic Affairs
Locations (1):
- Scripps Clinic at Torrey Pines, La Jolla, California, United States

REFERENCES:
- [Background] Stevenson DD. Aspirin desensitization in patients with AERD. Clin Rev Allergy Immunol. 2003 Apr;24(2):159-68. doi: 10.1385/CRIAI:24:2:159. PMID 12668896
- [Background] Berges-Gimeno MP, Simon RA, Stevenson DD. Long-term treatment with aspirin desensitization in asthmatic patients with aspirin-exacerbated respiratory disease. J Allergy Clin Immunol. 2003 Jan;111(1):180-6. doi: 10.1067/mai.2003.7. PMID 12532116